CLINICAL TRIAL: NCT05258487
Title: The Utility of the Validated Intraoperative Bleeding Scale in Spine Surgery
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Steven Ludwig, Chief of Spine Surgery, Professor, University of Maryland, Baltimore
Other Study IDs: HP-00097392
Record Dates: First submitted 2022-02-07; First posted 2022-02-28 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Intraoperative Blood Loss; Thoracolumbar Spine Surgery
Keywords: Blood Loss; Thoracolumbar Spine Surgery; VIBe; Blood Transfusion
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- VIBe Grade 1: Intraoperative bleeding of grade 1 as defined by the VIBe scale.
- VIBe Grade 2: Intraoperative bleeding of grade 2 as defined by the VIBe scale.
- VIBe Grade 3: Intraoperative bleeding of grade 3 as defined by the VIBe scale.
- VIBe Grade 4: Intraoperative bleeding of grade 4 as defined by the VIBe scale.

SUMMARY:
This is a single-center, prospective, observational study that will compare the blood transfusion rate between intraoperative bleeding severity characterized using the Validated Intraoperative Bleeding Scale (VIBe).

DETAILED DESCRIPTION:
Primary Aim: Assess the association between the VIBe scale and intraoperative and postoperative blood transfusion rates for posterior thoracolumbar spine surgery.

Primary Hypothesis: Patients with higher recorded VIBe grades during the five stages of spine surgery (exposure, decompression, instrumentation, fusion, and closing) will have a higher rate of receiving blood transfusions.

Secondary Aims: Determine the association between the VIBe scale and other postoperative outcomes and complications.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 88 years
* Patients receiving elective open, posterior thoracolumbar surgery

Exclusion Criteria:

* Patients receiving non-elective or trauma surgery
* Patients with pathologic spine fracture or metastatic disease to the spine
* Patients receiving thoracolumbar surgery through anterior or lateral approach
* Patients receiving spine surgery for debridement of suspected or confirmed infection

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective open, posterior thoracolumbar surgery
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Receiving Perioperative Blood Transfusion | From day of surgery until discharge from hospital, assessed up to 2 weeks following surgery.
  The main outcome will be whether or not the patient received a blood transfusion during the surgery or the postoperative hospitalization period.

SECONDARY OUTCOMES:
Total Estimated Blood Loss During Surgery (mL) | From the start to the end of surgery, assessed up to 1 day following surgery when estimated blood loss is reported and documented.
  The secondary outcome will be total blood loss during surgery assessed using anesthesiology and surgeon reported estimated blood loss (mL).

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Ludwig, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewis KM, Li Q, Jones DS, Corrales JD, Du H, Spiess PE, Lo Menzo E, DeAnda A Jr. Development and validation of an intraoperative bleeding severity scale for use in clinical studies of hemostatic agents. Surgery. 2017 Mar;161(3):771-781. doi: 10.1016/j.surg.2016.09.022. Epub 2016 Nov 10. PMID 27839931